CLINICAL TRIAL: NCT02671071
Title: Prospective Evaluation of Patients With Uterine Cervical Cancer in Brazilian Health Institutions - The EVITA I Study
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: EVA - Grupo Brasileiro de Tumores Ginecológicos (Unknown); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 0215/EVA 001
Record Dates: First submitted 2016-01-15; First posted 2016-02-02 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Cervix Cancer
Keywords: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Quality of Life Questionnaire (QLQ) — The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Cervical cancer module (EORTC QLQ-CX24) will be applied to all patients at 0, 3, 6, 12, 24, 36 months.

SUMMARY:
The primary objective of this study is to describe the socio-demographic, clinical pathological, quality of life and treatment characteristics of patients diagnosed with CC in Brazil.

DETAILED DESCRIPTION:
The primary objective of this study is to describe the socio-demographic, clinical pathological, quality of life and treatment characteristics of patients diagnosed with cervix cancer (CC) in Brazil. Other specific objectives are:

* To describe socio-demographic characteristics: age at diagnosis, education, family income, race, occupation, personal health habits - e.g.oral contraceptive use ever/never and duration; smoking never/ever/current/duration , ever drinking), sexual history, insurance coverage (private, public), institution (private, public, philanthropic), obstetric history, comorbidities, performance status, human papillomavirus vaccination or not
* To describe the screening for CC: access, type, frequency and results.
* To describe clinical pathological characteristics of CC: histology (adeno x squamous x adenosquamous x neuroendocrine x other) , International Federation of Gynecology and Obstetrics (FIGO) stage, pathological stage, exams for staging, date of diagnosis, site of metastasis.
* To describe treatment characteristics of CC: date of surgery, type of surgery; date and duration of radiotherapy, type of radiotherapy; date, type and lines of systemic therapy (chemotherapy, monoclonal antibodies),
* To describe treatment safety (grade 3-4 AEs, death due to treatment toxicity, discontinuation due to AE). In addition adverse events of special interest will be described (details on Safety section).
* To describe the outcomes: follow-up exams and date of visits, persistent disease, recurrence, progression times in metastatic disease, complications (e.g. hydronephrosis/nephrostomy/ GI perforations and both GI & genitourinary fistulae.), death due CC and death from any cause.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmed invasive cervical cancer
* Diagnosis of FIGO stages
* Stage 1B to 2A high risk
* 2B-4B or recurrent disease
* Patients ≥18 years old

Exclusion Criteria:

1. Non-invasive uterine carcinoma;
2. Pregnancy;
3. synchronous tumor or second primary tumor in the past 5 years (except thyreoid ancer or non-melanoma skin cancer).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cervical cancer in 1-year period (recently diagnosed IB to IIA high risk or IIB-IVB or recurrent disease - FIGO stages) at the participating sites will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 638 (Actual)
Dates: Start 2016-04; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Characterization of cervix cancer in the Brazilian female population | 3 years

SECONDARY OUTCOMES:
Socio-demographic characteristics of the female population diagnosed with CC | Month 0 (beginning of the study)
Description of the method used to diagnose the brazillian female patients with cervix cancer | Month 0
  Screening tests (Papanicolaou test) or symptoms presented by patients
The clinical and pathological characteristics of cervix cancer in brazilian female patients | Month 0
Type of treatment assessed in patients with CC | Month 0, 3, 6,12, 24 and 36
  Radiotherapy, Chemotherapy and/or Surgery
Number of patients with disease survival | Month 3, 6, 12, 24 and 36
Number of patients with progression survival | Month 3, 6, 12, 24 and 36
Number of patients with overall survival | Month 3, 6, 12, 24 and 36
Number of patients with disease overall survival | Month 3, 6, 12, 24 and 36
Type and description of the indicated treatment after the diagnosis of cervix cancer in brazilian female patients | Month 0, 3, 6,12, 24 and 36
Duration of treatment after the diagnosis of cervix cancer | Month 0, 3, 6,12, 24 and 36
Description of adverse effects of the cervix cancer treatment | Month 0, 3, 6,12, 24 and 36
Number of adverse effects of the cervix cancer treatment | Month 0, 3, 6,12, 24 and 36
Type of clinical outcomes of the patients with cervix cancer in Brazil | Month 0, 3, 6,12, 24 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group
Locations (16):
- Brazil (16):
  - Fundação Centro de Controle do Câncer do Estado do Amazonas, Manaus, Amazonas
  - CRIO, Fortaleza, Ceará
  - Clínica AMO, Salvador, Estado de Bahia
  - HU Walter Cantídeo, Ceará, Fortaleza
  - Hospital Alderona Bello, São Luís, Maranhão
  - UFMG, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - IMIP, Recife, Pernambuco
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - CPO - Hsl/Pucrs, Porto Alegre, Rio Grande do Sul
  - Hospital Geral de Roraima, Boa Vista, Roraima
  - CEPON, Florianópolis, Santa Catarina
  - Centro de Novos Tratamentos Litoral - Itajaí, Itajaí, Santa Catarina
  - INCA, Rio de Janeiro
  - Hospital São José, São Paulo
  - Instituto Brasileiro de Controle do Câncer - IBCC, São Paulo

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Munoz N, Franco EL, Herrero R, Andrus JK, de Quadros C, Goldie SJ, Bosch FX. Recommendations for cervical cancer prevention in Latin America and the Caribbean. Vaccine. 2008 Aug 19;26 Suppl 11:L96-L107. doi: 10.1016/j.vaccine.2008.05.062. PMID 18945407
- [Background] Hellner K, Munger K. Human papillomaviruses as therapeutic targets in human cancer. J Clin Oncol. 2011 May 1;29(13):1785-94. doi: 10.1200/JCO.2010.28.2186. Epub 2011 Jan 10. PMID 21220591
- [Background] Martinez-Mesa J, Werutsky G, Campani RB, Wehrmeister FC, Barrios CH. Inequalities in Pap smear screening for cervical cancer in Brazil. Prev Med. 2013 Oct;57(4):366-71. doi: 10.1016/j.ypmed.2013.06.026. Epub 2013 Jul 1. PMID 23827721
- [Background] Zuliani AC, Esteves SC, Teixeira LC, Teixeira JC, de Souza GA, Sarian LO. Concomitant cisplatin plus radiotherapy and high-dose-rate brachytherapy versus radiotherapy alone for stage IIIB epidermoid cervical cancer: a randomized controlled trial. J Clin Oncol. 2014 Feb 20;32(6):542-7. doi: 10.1200/JCO.2013.50.1205. Epub 2014 Jan 21. PMID 24449243
- [Background] Pearcey R, Brundage M, Drouin P, Jeffrey J, Johnston D, Lukka H, MacLean G, Souhami L, Stuart G, Tu D. Phase III trial comparing radical radiotherapy with and without cisplatin chemotherapy in patients with advanced squamous cell cancer of the cervix. J Clin Oncol. 2002 Feb 15;20(4):966-72. doi: 10.1200/JCO.2002.20.4.966. PMID 11844818